CLINICAL TRIAL: NCT00901368
Title: A PHASE 4, MULTINATIONAL, MULTICENTRE, DOUBLE BLIND, DOUBLE DUMMY, RANDOMIZED, PARALLEL GROUP, CONTROLLED CLINICAL STUDY OF FIXED COMBINATION BECLOMETHASONE DIPROPIONATE 100 µg PLUS FORMOTEROL FUMARATE 6 µg pMDI WITH HFA-134A PROPELLANT (CHF1535, FOSTER®) VERSUS FLUTICASONE 250 µg PLUS SALMETEROL 50 µg DPI (SERETIDE® DISKUS®) AS MAINTENANCE TREATMENT IN CONTROLLED ASTHMATIC PATIENTS.
Brief Title: FACTO Study (Foster® As Complete Treatment Option)
Acronym: FACTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-0806-PR-0032; 2008-003740-11 (EudraCT Number)
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthmatic Patients
MeSH Terms: interventions — Foster Home Care; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CHF1535 (beclometasone dipropionate plus formoterol, 400/24 µg daily)
  Interventions: Drug: FOSTER
- 2 (Active Comparator): Seretide® Diskus® (fluticasone plus salmeterol, 500/100 µg /daily)
  Interventions: Drug: Seretide

INTERVENTIONS:
Drug: FOSTER — CHF1535 (beclometasone dipropionate 100 µg plus formoterol 6 µg) pMDI aerosol via HFA-134a propellant 2 inhalations b.i.d. (daily dose 400 µg + 24µg)
  Arms: 1
Drug: Seretide — Fluticasone 250 µg + salmeterol 50 µg DPI (Seretide® Diskus®) 1 inhalation b.i.d. (daily dose 500+100 µg)
  Arms: 2

SUMMARY:
Double blind, multinational, multicentre, randomised, 2 arm parallel group study

DETAILED DESCRIPTION:
Aim of the present investigation is to demonstrate the clinical equivalence between fluticasone plus salmeterol 500/100 µg daily and an equipotent dose of CHF1535 in maintaining the same asthma control in patients adequately controlled with fluticasone plus salmeterol at the above mentioned daily dose.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic patients will be enrolled at Visit 1 into the run-in period if they meet all of the following criteria:

1. Written informed consent obtained
2. Adult male and female (≥18 and ≤65 years)
3. Clinical diagnosis of controlled asthma according to Global Strategy for Asthma Management and Prevention (GINA) revised version 2007 in the previous week before study entry:

   * no daytime symptoms (twice or less/week)
   * no limitations of activities
   * no nocturnal symptoms/awakenings
   * no need for reliever/rescue medications (twice or less/week)
   * lung function (FEV1) > 80% predicted or personal best (if known)
4. Patients treated with fluticasone 500 µg + salmeterol 100 µg daily for ≥ 4 weeks
5. A co-operative attitude and ability to correctly use the device and to complete the diary cards.

Exclusion Criteria:

Patients will not be enrolled at visit 1 into the run-in period if they meet any of the following criteria:

1. Inability to carry out pulmonary function testing;
2. Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the National Heart Lung and Blood Institute/World Health Organisation (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines;
3. History of near fatal asthma;
4. Evidence of severe asthma exacerbation or symptomatic infection of the lower airways in the previous six months;
5. Three or more courses of oral corticosteroids or hospitalisation due to asthma during the previous 6 months;
6. Patients treated with long-acting β2-agonists (LABAs) other than salmeterol, anticholinergics, and leukotriene antagonists during the previous 4 weeks;
7. Current smokers or recent (less than one year) ex-smokers defined as smoking at least 15 packs/year;
8. Clinically significant or unstable concurrent disease : e.g. uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; significant other pulmonary disease; cardiovascular disease; gastrointestinal disease; neurological disease; haematological disease, autoimmune disorders, that may interfere with patient's safety, compliance, or study evaluations, according to the investigator's opinion;
9. Patients with a serum potassium value ≤ 3.5 mEq/L
10. Patients with QTc interval (Bazett's formula) higher than 450 msec at screening visit 1;
11. Cancer or any chronic diseases with prognosis < 2 years;
12. Female subjects: pregnant or with active desire to be pregnant, lactating mother or lack of efficient contraception in a subject with child-bearing potential (i.e. contraceptive methods other than oral contraceptives, IUD, tubal ligature). A pregnancy test in urine is to be carried out in women of a fertile age at screening
13. Significant alcohol consumption or drug abuse;
14. Patients treated with beta-blockers as regular use;
15. Patients treated with monoamine oxidase inhibitor, tricyclic antidepressants and Selective Serotonin Re-uptake Inhibitors (SSRIs), unless already taken at stable doses at the screening visit
16. Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
17. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
18. Patients who received any investigational new drug within the last 12 weeks;
19. Patients with asthma exacerbations during the run-in period will also be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pre-dose morning FEV1 measured at clinic visit 5 | 12-week treatment

SECONDARY OUTCOMES:
FEV1 area under the curve (AUC) in the first hour post-dose measured at clinics at visit 2 and visit 5 | 12-week treatment
Pulmonary function tests measured at clinics (FEV1,PEF, FVC, FEF25-75%) | 12-week treatment
ACQ score at baseline and at the end of treatment period | 12-week treatment
Use of rescue medication | 12-week treatment
Number of patients with controlled or partly controlled asthma at clinic visits according to GINA guidelines revised version 2007 | 12-week treatment
Days without asthma symptoms (%), days without use of rescue medication (%) and daily asthma symptoms' score from diary cards | 12-week treatment
Pharmacoeconomic analyses assessing differences in direct medical costs (healthcare perspective) and in both direct healthcare and indirect costs (societal perspective). | 12-week treatment
Adverse events and adverse drug reactions,ECG ,Vital signs, Haematology/blood chemistry tests, OUCC ratio in a in a subgroup of 15% of patients | 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neil Barnes, MD, Principal Investigator — Department ofRespiratory Medicine, London Chest Hospital, Barts& The London NHS Trust,Bonner Road, E2 9JX, London (UK)
Locations (4):
- Hôpital Nord, Marseille, France
- Allergologie imUmkreis der Praxis Pneumologie, Gelsenkirchen, North Rhine-Westphalia, Germany
- Atrium Medisch Centrum Heerlen,, Heerlen, Netherlands
- Hospital Universitario La Fe, Valencia, Spain

REFERENCES:
- [Result] Barnes N, van Noord JA, Brindicci C, Lindemann L, Varoli G, Perpina M, Guastalla D, Casula D, Patel S, Chanez P; FACTO (Foster(R) As Complete Treatment Option) Study Group. Stepping-across controlled asthmatic patients to extrafine beclometasone/formoterol combination. Pulm Pharmacol Ther. 2013 Oct;26(5):555-61. doi: 10.1016/j.pupt.2013.01.011. Epub 2013 Mar 22. PMID 23524015
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2008-003740-11